### **SEMMELWEIS UNIVERSITY**

Department of Vascular Surgery and Endovascular Therapy
Head of Department: Dr. Péter Sótonyi
Address: 1122 Budapest, Városmajor u. 68.
E-mail: titkarsag.erseb@semmelweis-univ.hu
Tel.: (+36-1) 458-6795

## STUDY DOCUMENT COVER PAGE

### Official Title of the Study

"Local and systemic immune and inflammatory protective mechanisms and risk factors in the progression of carotid artery stenosis and aortic aneurysm"

### **ClinicalTrials.gov Identifier (NCT Number)**

Not yet assigned

# **Type of Document**

Patient Informed Consent Form

**Date of Document** 

2025-10-1

Version

Version [1.1]



#### SEMMELWEIS UNIVERSITY

Department of Vascular and Endovascular Surgery

Head of Department Dr. Péter Sótonyi

Patient Declaration on Participation in the Research Study Titled 'Local and Systemic Immune - and Inflammatory Protective Mechanisms and Risk Factors in the Progression of Carotid Artery Stenosis and Aortic Aneurysm' I hereby consent to participate in

| clinical investigation conducted by<br>Department of Vascular Surgery a | Ind Endovascular The nt and detailed information in the second ask my que had sufficient time to my intention to particular any coercion. | erapy, Városmajor Heart and Vas-<br>nation concerning the microbiome-<br>uestions and that I received satis-<br>to read and comprehend the<br>icipate in the study. I have made<br>I understand that I may withdraw | e |
|---|---|---|---|
| Participant in the study: | | | |
| Name: | | | |
| Mother's name: | | | |
| Place and date of birth:<br>Address: | | | |
| Signature of the study participant | | <br>Date | |
| Declaration of the investigating | nhysician | | |
| By signing this declaration, I hereby confi<br>prehensive and thorough information abo<br>that the patient clearly understood the na | rm that, to the best of my<br>out the study at the time o | of signing the informed consent, and | |
| Physician's name, registration number | | Physician's signature | |

Thank you for your cooperation.

